CLINICAL TRIAL: NCT04672330
Title: A Phase II Study of Tislelizumab(T) as Neoadjuvant Treatment for Cisplatin-ineligible High Risk Upper Tract Urothelial Carcinoma (UTUC)
Brief Title: Neoadjuvant PD-1 Monoclonal Antibody in Cisplatin-ineligible High Risk Upper Tract Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO-IO
Record Dates: First submitted 2020-12-12; First posted 2020-12-17 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Neoadjuvant Immunotherapy of Cisplatin-ineligible High Risk Upper Urinary Tract Urothelial Carcinoma
Keywords: neoadjuvant therapy; radical nephroureterectomy; Tislelizumab; Cisplatin-ineligible
MeSH Terms: interventions — tislelizumab; spartalizumab

STUDY DESIGN:
Intervention Model Description: Patients will receive 2-4 cycles of Tislelizumab (200mg per cycle) prior to surgery（radical nephroureterectomy, segmental ureteral resection, endoscopic ablation）
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant arm (Experimental): Patients will receive 2-4 cycles of Tislelizumab (200mg per cycle) prior to surgery（radical nephroureterectomy, segmental ureteral resection, endoscopic ablation） Drug: Tislelizumab 200 mg per cycle, IV on day 1 of every 3-week cycle, for 2-4 cycles prior to surgery
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Patients will receive 2-4 cycles of Tislelizumab (200mg per cycle) before surgery（radical nephroureterectomy, segmental ureteral resection, endoscopic ablation）
  Other Names: anti-PD-1 monoclonal antibody

SUMMARY:
Neoadjuvant therapy of cisplatin-based chemotherapy has been proved to improve prognosis of muscle invasive UTUC patients in several studies. This study is designed to investigate the safety and efficacy of neoadjuvant PD-1 monoclonal antibody in patients with locally advanced upper urinary tract urothelial carcinoma (UTUC) which are ineligible for cisplatin. Tislelizumab, an anti-programmed death protein-1 (PD-1) monoclonal antibody, was engineered to minimize binding to FcγR on macrophages to abrogate antibody-dependent phagocytosis, a mechanism of T-cell clearance and potential resistance to anti-PD-1 therapy. The safety, tolerability, and efficacy of tislelizumab in patients with PD-L1 positive urothelial carcinoma who progressed during/following platinum-containing therapy was proved in a phase 2 trial (CTR20170071). This trial focuses on the efficacy of Tislelizumab to induce pathological down-staging of locally advanced UTUC in neoadjuvant setting.

DETAILED DESCRIPTION:
Neoadjuvant therapy of cisplatin-based chemotherapy has been proved to improve prognosis of muscle invasive UTUC patients in several studies. This study is designed to investigate the safety and efficacy of neoadjuvant PD-1 monoclonal antibody in patients with locally advanced upper urinary tract urothelial carcinoma (UTUC) which are ineligible for cisplatin. Tislelizumab, an anti-programmed death protein-1 (PD-1) monoclonal antibody, was engineered to minimize binding to FcγR on macrophages to abrogate antibody-dependent phagocytosis, a mechanism of T-cell clearance and potential resistance to anti-PD-1 therapy. The safety, tolerability, and efficacy of tislelizumab in patients with PD-L1 positive urothelial carcinoma who progressed during/following platinum-containing therapy was proved in a phase 2 trial (CTR20170071). This trial focuses on the efficacy of Tislelizumab to induce pathological down-staging of locally advanced UTUC in neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* 1. had non-metastatic high risk UTUC and planed to receive surgery(defined as high grade UTUC either by endoscopic biopsy or urinary cytology and/or any invasive aspect on radiological examination and/or hydronephrosis );
* 2. were ineligible for cisplatin-based chemotherapy(defined as meeting at least one of the following criteria: Eastern Cooperative Oncology Group [ECOG] performance status 2, creatinine clearance 30-60 mL/min, grade ≥2 audiometric hearing loss, grade ≥2 peripheral neuropathy, or New York Heart Association Class III heart failure);
* 3. had not received any systemic anti-tumor therapy;
* 4. Adequate organ function defined by study-specified laboratory tests; Hemoglobin ≥90 g/L; Hematological Absolute neutrophil count (ANC) ≥1.5×109 /L; Platelets ≥100×109 /L
* 5. No functional organic disease: T-BIL≤1.5×upper limit of normal (ULN); ALT andAST≤2.5×ULN; Serum creatinine≤2×ULN; endogenous creatinine clearance rate>30ml/min
* 6. Agree to comply with scheduled visits, treatment plans, lab tests and any other required study procedures;

Exclusion Criteria:

* 1. Patients who have received prior therapy of an anti-PD-1, anti-PD-L1, or anti-PD-L2 antibody;
* 2. Patients who are allergic to monoclonal antibodies or any of its excipients;
* 3. Patients who have received other systems for anti-tumor treatment (e. g., Steroid therapy, immunotherapy) within 4 weeks or enrolled in other clinical trials;
* 4. Patients who are pregnant or breastfeeding, or expecting to conceive;
* 5. Patients who have a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies);
* 6. Patients who have known active Hepatitis B or Hepatitis C;
* 7. Patients who have active autoimmune disease that has required systemic treatment in the past 2 years;
* 8. Patients who have received a live vaccine within 30 days prior to the first dose of trial treatment;
* 9. Patients who have received prior radiation therapy to the bladder;
* 10.Patients who have muscle invasive bladder cancer;
* 11.Patients who have received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
* 12.Patients who have a history of substance abuse or with a history of mental disorders;
* 13.Patients who had other malignant tumors in the past five years that have not recovered except for curable tumors that have been cured including basal or squamous skin cancer, localized carcinoma in situ of the cervix or the breast and low-risk prostate cancer, etc.
* 14.Patients who have active tuberculosis;
* 15.Patients who have other serious and uncontrollable accompanying diseases that may affect compliance or interfere with the interpretation of results including active opportunistic infections or advanced (severe) infections, uncontrollable diabetes, cardiovascular disease (grade III or IV heart failure defined by the New York Heart Association classification, II degree atrioventricular block and above, myocardial infarction in the past 6 months, unstable arrhythmia or instability angina, cerebral infarction within 3 months, etc.) or lung disease (interstitial pneumonia, history of obstructive lung disease and symptomatic bronchospasm);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
pathological reponse rate | 30 days after surgery
  ypT0N0 at surgical specimen，in the intention-to-treat population

SECONDARY OUTCOMES:
pathological response rate | 30 days after surgery
  ypT0 and ypT1 at surgical specimen，in the intention-to-treat population
perioperative complication rate | 30 days after surgery
  the rate of perioperative complications are determined according to Clavien classification
objective response rate | 12 months after drug treatment
  the proportion of patients with a confirmed complete response or partial response based on radiological examination before surgery per RECIST version 1.1
disease free survival | 5 years after surgery or treatment
  from surgery to any kind of recurrence including tumour bed, first metastasis, or death from any cause
overall survival | 5 years after enrollment
  time from enrollment to death for any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang J, Cai X, Ng C, Luo Y, Chen Q, Wang Z, Qiao K, Kong W, Zhang J, Chen Y, Zhang W, Zhang J, Zhang D, Wu G, Chen H, Xue W. A Phase 2 Study of Tislelizumab as Neoadjuvant Treatment of Cisplatin-Ineligible High-Risk Upper Tract Urothelial Carcinoma. J Urol. 2025 Jun;213(6):739-752. doi: 10.1097/JU.0000000000004475. Epub 2025 Feb 25. PMID 39999445